CLINICAL TRIAL: NCT00451542
Title: Time to Relapse During Treatment With Divalproex vs. Lamotrigine for Bipolar Disorder
Brief Title: Divalproex vs. Lamotrigine for Bipolar Disorder
Status: Terminated | Type: Observational
Why Stopped: Sample too small in retrospective chart review to conduct analysis
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Responsible Party: Principal Investigator, Lori Davis, MD, ACSO R&D, Tuscaloosa Research & Education Advancement Corporation
Other Study IDs: 0063
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Relapse; Retrospective
MeSH Terms: conditions — Bipolar Disorder; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective chart review of patients treated for bipolar disorder at the TVAMC in the past four years cross-referenced with the electronic pharmacy file for having received a prescription of divalproex or lamotrigine.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the long-term outcome in bipolar patients treated with divalproex versus lamotrigine in a retrospective chart review of veterans as measured by time to relapse into any significant mood episode (i.e. mania or depression). The primary hypothesis is that bipolar patients will demonstrate significantly greater time to relapse in those treated with divalproex compared to those treated with lamotrigine. The secondary objective of the study is to assess the safety and relative tolerability of divalproex and lamotrigine in this population based on discontinuation due to side or adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar I or Bipolar II disorder
* Prescription of divalproex (any formulation except for Depakene/valproic acid) or lamotrigine in the electronic pharmacy profile.
* Age 19 or older
* Demonstrated stability for at least 4 weeks on an adequate dose of each medication (at least 50mg/d lamotrigine or 15mg/kg/day divalproex).
* Treatment at the TVAMC for at least 6 months following the prescription of divalproex or lamotrigine.

Exclusion Criteria:

* Primary diagnosis of schizoaffective or schizophrenia during the evaluation period.
* Prescription of divalproex and lamotrigine given concurrently during the observation period.
* History of Dementia or cognitive disorders

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Bipolar Disorder I or II who had a prescription of divalproex or lamotrigine.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2008-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Reseach and Education Advancement Corporation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vieta E, Rosa AR. Evolving trends in the long-term treatment of bipolar disorder. World J Biol Psychiatry. 2007;8(1):4-11. doi: 10.1080/15622970601083280. PMID 17366344